CLINICAL TRIAL: NCT05270590
Title: Early Outcome of Minimally Invasive Rheumatic Mitral Valve Surgery Through Periareolar Versus Submamary Approach
Brief Title: Minimally Invasive Rheumatic Mitral Valve Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Rabee Hamed Ahmed, assistant lecture at cardiothoracic department, Assiut University
Other Study IDs: peri areolar MVR
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Rheumatic Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: periareolar approach
  Interventions: Procedure: minimally invasive rheumatic mitral valve surgery
- group B: submamary approach
  Interventions: Procedure: minimally invasive rheumatic mitral valve surgery

INTERVENTIONS:
Procedure: minimally invasive rheumatic mitral valve surgery — First, venous and arterial access was established. Incision establishment: A 4 to 6 cm incision was opened in the chest anterolaterally to the right of the fourth intercostal space (in submamarry vs. peri areolar approach ). The thoracoscope was inserted. Bypass started, and Chitwood occlusion forceps were inserted to block the ascending aorta, purse-string suturing of the cardioplegia cannula and antegradecardioplegia fluid was performed, the interatrial groove was freed, the left atrial incision was made. Removal of the damaged mitral valve mostly by endoscopic surgical instruments (not usually there is a chance for repair), and the mitral valve was sutured intermittently. After examination of the valve location and the opening and closing performance of the valve leaf, the left atrial incision was sutured continuously by prolene 4/0. Weaning from bypass start

SUMMARY:
Early outcome of minimally invasive rheumatic mitral valve surgery through periareolar versus submamary approach

DETAILED DESCRIPTION:
Rheumatic heart valve disease (RHVD) is a post-infectious sequel of acute rheumatic fever resulting from an abnormal immune response to a streptococcal pharyngitis that triggers valvular damage. RHVD is the leading cause of cardiovascular death in children and young adults, mainly in women from low and middle-income countries. It is known that long-term inflammation and high degree of fibrosis leads to valve dysfunction due to anatomic disruption of the valve apparatus.in low and middle-income countries, rheumatic heart valve disease (RHVD) is the leading cause of cardiovascular death in children and young adults When there is severe valvular dysfunction, especially if the patient is symptomatic, surgery is indicated. (1)Traditional mitral valve surgery via a median sternotomy is safe and effective, but it results in a high degree of trauma and a long incision.(2) In the last 2 decades, a minimally invasive (MI) technique has been used widely in cardiac surgery.(3-4) Its prominent advantage in post-surgery recovery and the small incision required makes patients prefer it over a traditional incision.(5-6) Patients underwent Minimal invasive surgery after intravenous anaesthesia combined with general anaesthesia, and their right side was elevated at 30°. After disinfection and draping were performed with sterile protective film fixed to it. Establishing the in vitro pathway: First, venous and arterial access was established. Incision establishment: A 4 to 6 cm incision was opened layer by layer in the chest anterolaterally to the right of the fourth intercostal space (in submamarry vs. peri areolar approach ). A lap-protector was placed. The thoracoscope was inserted near the anterior axillary line of the third intercostal space into the chest with CO2 input. A pericardial longitudinal incision was made under direct vision, extending to the head side and reflexed when reaching the aorta, with the pericardium suspended. Extracorporeal circulation was started, and Chitwood occlusion forceps were inserted into the chest to block the ascending aorta through the fourth intercostal space; the drainage tube of the left atrium perforated the chest through the right midaxillary line between the fifth and sixth intercostal space. 4-0 Prolene was used for the purse-string suturing of the cardioplegia cannula and antegradecardioplegia fluid was performed. After electrocardiograph monitoring showed that electrocardiac activity had stopped, the interatrial groove was freed, the left atrial incision was made parallel to the interatrial groove, and the left atrial drainage tube was inserted. A left atrial retractor was placed and stretched to the surface for fixation through the perforation into the prothorax, and the left atrial incision was retracted in the direction of the sternum. Removal of the damaged mitral valve by endoscopic surgical instruments, and the mitral valve was sutured intermittently. After examination of the valve location and the opening and closing performance of the valve leaf, the left atrial incision was sutured continuously by prolene 4/0. Retrograde cardioplegia perfusion through the tube was initiated for venting and rewarming of the patient started, and the anesthesiologist ventilated the lungs with air to keep the lung lobes full and to relieve the occlusion of the ascending aorta. Cardiopulmonary bypass was stopped gradually and bleeding was stopped; a chest drainage tube was inserted through the hole for the left atrium drainage tube, and the chest was closed.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of rheumatic mitral valve
2. Patient undergoing minimal invasive rheumatic mitral valve surgery
3. Patient is willing to comply with all follow-up visits.
4. Willing and able to provide written informed consent and comply with study requirements

Exclusion Criteria:

1. Ischemic heart disease
2. Patients need another valve replacement
3. Redo mitral valve replacement

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patient undergoing minimal invasive rheumatic mitral valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
identify of advantages and disadvantages of each approach | 1/1/2022 TO 1/1/2025
  discussing and finding each approachs advantages and disadvantages and comparing with each other
Assess the outcome regarding: -Wound size | 1/1/2022 TO 1/1/2025
  measuring Wound size (in cm ) of each approach
Assess the outcome regarding: -Postoperative pain and patient satisfaction | 1/1/2022 TO 1/1/2025
  measuring postoperative pain and patient satisfaction by pain scale of each approach
assess Wound complication | 1/1/2022 TO 1/1/2025
  assess Wound complication (as infection (superfacial , deep , burst chest )

SECONDARY OUTCOMES:
Assess the outcome regarding: Economic factor | 1/1/2022 TO 1/1/2025
  Assess the outcome regarding:
  -Economic factor ( ICU stay or hospital stay)
Assess the outcome regarding:Time of procedure | 1/1/2022 TO 1/1/2025
  Assess the outcome regarding:Time of procedure ( time of total bypass time , time for rapid access, time of haemostasis)

CONTACTS AND LOCATIONS:
Overall Officials: Anwar A Atia, MD in cardiothoracic surgery, Study Chair — Professor of cardiothoracic surgery; Ahmed N Malik, MD in cardiothoracic surgery, Study Chair — Professor of cardiothoracic surgery

REFERENCES:
- [Background] Watkins DA, Johnson CO, Colquhoun SM, Karthikeyan G, Beaton A, Bukhman G, Forouzanfar MH, Longenecker CT, Mayosi BM, Mensah GA, Nascimento BR, Ribeiro ALP, Sable CA, Steer AC, Naghavi M, Mokdad AH, Murray CJL, Vos T, Carapetis JR, Roth GA. Global, Regional, and National Burden of Rheumatic Heart Disease, 1990-2015. N Engl J Med. 2017 Aug 24;377(8):713-722. doi: 10.1056/NEJMoa1603693. PMID 28834488
- [Background] Antunes MJ. Minimally invasive valve surgery: reality, dream or utopia? J Heart Valve Dis. 1998 Jul;7(4):358-9. No abstract available. PMID 9697053
- [Background] Takeda M, Konishi T, Fukata M, Matsuzaki K, Furuya K. [Minimally invasive surgery for single valvular heart disease]. J Cardiol. 1999 Oct;34(4):219-23. Japanese. PMID 10553539
- [Background] Modi P, Hassan A, Chitwood WR Jr. Minimally invasive mitral valve surgery: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2008 Nov;34(5):943-52. doi: 10.1016/j.ejcts.2008.07.057. Epub 2008 Sep 30. PMID 18829343